CLINICAL TRIAL: NCT06112886
Title: Identification of Important Symptoms and Diagnostic Hypothyroidism Patients Using Machine Learning Algorithms
Status: Completed | Type: Observational
Sponsor: Kerman University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Salahodin rakhshani rad, Principal Investigator, Kerman University of Medical Sciences
Other Study IDs: 401000292
Record Dates: First submitted 2023-10-25; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Prediction Hypothyroidism Patients Using Machine Learning Algorithms; Identification of Important Symptoms of Hypothyroidism
Keywords: Hypothyroidism; Machine learning algorithms; Random Forest; Decision tree; Logistic regression
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- with Hypothyroidism, without Hypothyroidism
  Interventions: Other: There was no intervention in this study

INTERVENTIONS:
Other: There was no intervention in this study — There was no intervention in this study

SUMMARY:
Hypothyroidism (HT) is one of the most common endocrine diseases. It is, however, usually challenging for physicians to diagnose due to non-specific symptoms. The usual procedure for diagnosis of HT is a blood test. In recent years, machine learning algorithms have proved to be powerful tools in medicine due to their diagnostic accuracy. In this study, we aim to predict and identify the most important symptoms of HT using machine learning algorithms.

DETAILED DESCRIPTION:
Hypothyroidism (HT) is one of the most common diseases in the world, in which insufficient thyroid hormone is produced. Due to the wide variation in clinical symptoms, the definition of HT is mainly biochemical. Ninety nine percent of primary cases of HT are related to deficiency of thyroxine (T4) and triiodothyronine (T3) hormones. Deficiency in T4 and T3 hormones, which are produced by thyroid gland, leads to increasing thyroid-stimulating hormone (TSH) production through a negative feedback mechanism .

HT has non-specific symptoms such as weight gain, fatigue, insufficient concentration, depression, menstrual irregularities, and constipation, which change with age, gender, and other factors. Autoimmune thyroiditis (Hashimoto's disease) is the most common symptom of this disorder.

The prevalence of HT is 2% in the world, even in the existence of enough iodine in daily food. In a cohort study that was conducted in Iran in 2017, a significant increase in the prevalence of thyroid dysfunction was reported, from 1.4 to 10.5, attributed to several factors such as geographical areas, aging, ethnicity and the amount of iodine intake.

Increasing in serum cholesterol levels and the risk of coronary artery disease and cardiovascular mortality are the most common complications of HT. The economic burden of HT is fairly high, especially in patients with other underlying diseases such as diabetes and hemodialysis. The common clinical method for diagnosing equally primary HT is to check the serum concentration of TSH; People with TSH and T4 levels above the reference age range are diagnosed as hypothyroid. The upper limit of the TSH reference range usually increases with age in adults .

In recent years, artificial intelligence and machine learning techniques have attracted increasing attention from medical researchers. Among the most attractive features of machine learning in medicine are disease prediction and diagnosis of simple symptoms . The prediction models such as support vector machine (SVM), decision tree (DT), random forest (RF) and artificial neural network (ANN), are among the most popular machine learning methods.

As accurate diagnostic of HT is currently based on the TSH level obtained by a blood test, it creates some expense burden and anxiety for patients. The aim of the present study is to first diagnose HT in new cases that have no history of HT symptoms with three statistical machine learning methods (logistic regression, decision tree and random forest). The diagnosis is performed using simple and widely-accepted visual symptoms of HT that endocrinologists identify. Second, the most important visual features of HT which can help physicians in diagnosis, are also ranked using decision tree and random forest methods.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hypothyroidism Disease
* aged 18 years or more

Exclusion Criteria:

* Having history of Hypothyroidism treatment and thyroid gland surgery
* Having HT during previous pregnancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The sexual identity of people is based on their physiological appearance
Study Population: In total 1296 individuals (1088 women and 208 men) aged 18 years or over participated in this cross-sectional study from September to December 2022 at our main clinic for thyroid treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1296 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
physiological parameter | 6 months
  Information about hypothyroidism was collected by checklist. Then, TSH test was used for each individual to obtain the response variable. People whose TSH level is above 4 mIU/L are identified as hypothyroid. A person whose TSH is between 0.4 and 0.4 mIU/L is considered healthy.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health, Kerman University of Medical Sciences, Kerman, Iran

IPD SHARING:
Plan to Share IPD: Yes
The data is related to the common symptoms of hypothyroidism. Also, this data includes 6 demographic variables. If a researcher conducts research on hypothyroidism and machine learning, he/she can access the data by citing sufficient reasons.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As soon as satisfactory confirmation is given, the data will be sent. This may take between one and two weeks
Access Criteria: Any research related to hypothyroidism and its diagnosis methods using simple symptoms. Use in the field of machine learning